CLINICAL TRIAL: NCT01479530
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study of [Azilect®] Rasagiline in Levodopa-treated Parkinson's Patients With Motor Fluctuations in China
Brief Title: Azilect® (Rasagiline) in Levodopa-treated Parkinson's Patients With Motor Fluctuations in China
Acronym: CHORAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13445A
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Rasagiline; Azilect; Parkinson´s Disease; Motor fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Azilect® (Experimental)
  Interventions: Drug: Azilect®

INTERVENTIONS:
Drug: Placebo — Once daily; tablet; orally; 16 weeks
  Arms: Placebo
Drug: Azilect® — 1 mg daily; tablet; orally; 16 weeks
  Other Names: Rasagiline
  Arms: Azilect®

SUMMARY:
The rationale for conducting this study is to evaluate the efficacy, tolerability, and safety of rasagiline compared to placebo in levodopa-treated Parkinson's Disease (PD) Chinese patients with motor fluctuations. Azilect® (Rasagiline) is indicated for the treatment of idiopathic PD as monotherapy (without levodopa) or as adjunct therapy (with levodopa) in patients with end of dose fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD.
* Patients with motor fluctuations averaging at least 1 hour daily in the "OFF" state during the waking hours.
* Patients with a Modified Hoehn and Yahr stage ≤3 in the "ON" state.
* Patients taking optimised levodopa or dopa decarboxylase inhibitor (DDI) therapy; they must be stable for at least 14 days prior to baseline.
* Patients receiving at least 3 daily doses of levodopa and not more than 8 daily doses of levodopa.
* Patients who have demonstrated the ability to keep accurate "24-hour" diaries prior to randomisation.

Exclusion Criteria:

* Patients with a clinically significant or unstable medical or surgical condition that would preclude his/her safe and complete study participation.
* Patients with a clinically significant or unstable vascular disease.
* Patients who have undergone a neurosurgical intervention of PD.
* Patients with severe disabling dyskinesias.
* Patients with a clinically significant psychiatric illness, including a major depression, which compromises their ability to provide consent or participate fully in the study.
* Patients with a Mini Mental State Examination (MMSE) score ≤24.
* Patients with a diagnosis of melanoma or a history of melanoma, or a suspicious lesion.

Other inclusion and exclusion criteria may apply.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (18):
- China (18):
  - CN015, Beijing
  - CN008, Beijing
  - CN017, Beijing
  - CN001, Beijing
  - CN018, Beijing
  - CN011, Chengdu
  - CN003, Guangzhou
  - CN005, Guangzhou
  - CN004, Hangzhou
  - CN019, Qingyu Zhou
  - CN020, Qingyu Zhou
  - CN012, Shanghai
  - CN007, Shanghai
  - CN013, Shanghai
  - CN006, Suzhou
  - CN009, Wuhan
  - CN010, Xi'an
  - CN014, Zi’an

REFERENCES:
- [Derived] Zhang Z, Shao M, Chen S, Liu C, Peng R, Li Y, Wang J, Zhu S, Qu Q, Zhang X, Chen H, Sun X, Wang Y, Sun S, Zhang B, Li J, Pan X, Zhao G. Adjunct rasagiline to treat Parkinson's disease with motor fluctuations: a randomized, double-blind study in China. Transl Neurodegener. 2018 Jun 30;7:14. doi: 10.1186/s40035-018-0119-7. eCollection 2018. PMID 29988514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients with a primary diagnosis of idiopathic Parkinson's disease.
Pre-assignment Details: The study consisted of a 2-week Screening Period during which the levodopa dose was optimised (if required), a 2-week Screening Period during which the levodopa dose was stabilised, a 16-week double-blind treatment period with rasagiline or placebo once daily (patients were randomised in a 1:1 ratio), and a 4-week Safety Follow-up Period.
Period: Overall Study
Arm/Group | Placebo | Azilect®
Started | 158 | 163
Completed | 148 | 151
Not Completed | 10 | 12
Not completed — Adverse Event | 5 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal of Consent | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azilect® | Total
Number analyzed (Participants) | 158 | 163 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] — all-patients-treated set (APTS) - all patients in the all-patients-randomised set (APRS) who took at least one dose of investigational medicinal product (IMP).
  years | 61.7 (9.9) | 62.7 (8.9) | 62.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants] — APTS
  Participants
    Female | 49 | 60 | 109
    Male | 109 | 103 | 212
Total Daily OFF Time [Mean (Standard Deviation); unit: hours] — Parkinson's Disease Patient Diary is a self-administered diary designed to assess motor fluctuations throughout the day. It is divided into 30-minute intervals, and the patient selects one of four options for each interval: asleep; off; on with no dyskinesia or without troublesome dyskinesia; or on with troublesome dyskinesia.
  Full-analysis set (FAS) - all patients in the APTS who had at least one valid post-baseline measurement of the total daily OFF time (a valid post-baseline diary was a diary reported from Week 4 onwards based on pre-defined visit windows).
  hours | 6.13 (2.72) | 6.10 (2.60) | 6.12 (2.66)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression - Severity of Illness (CGI-S) is a single-item rating scale used to evaluate a patient's severity of illness on a 7-point scale, based on the investigator's total clinical experience with patients. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  FAS.
  units on a scale | 4.07 (0.77) | 3.94 (0.76) | 4.00 (0.77)
UPDRS-ADL Score During OFF Time [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale (UPDRS) is a 42-item rating scale designed to assess PD-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worse outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: activities of daily living (ADL) - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
  FAS.
  units on a scale | 16.45 (7.54) | 15.59 (7.15) | 16.01 (7.34)
UPDRS Motor Score During ON time [Mean (Standard Deviation); unit: units on a scale] — UPDRS is a 42-item rating scale designed to assess PD-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worse outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: ADL - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
  FAS.
  units on a scale | 25.62 (10.48) | 23.82 (10.47) | 24.70 (10.50)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Total Daily OFF Time Using Parkinson's Disease Patient Diary
Description: Parkinson's Disease Patient Diary is a self-administered diary designed to assess motor fluctuations throughout the day. It is divided into 30-minute intervals, and the patient selects one of four options for each interval: asleep; off; on with no dyskinesia or without troublesome dyskinesia; or on with troublesome dyskinesia.
  The Change From Baseline in Mean Total Daily OFF time is calculated by taking the difference between the average of the total daily OFF time at Weeks 4, 8, 12, and 16, and the Baseline Total Daily OFF Time.
Time Frame: Baseline and Weeks 4, 8, 12, and 16
Population: Full-analysis set (FAS); observed cases (OC)
Measure: Mean (Standard Error); unit: hours
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 150 | 158
hours | -0.76 (0.16) | -1.25 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.0228, ANCOVA; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-0.92 to -0.07], Standard Error of Mean 0.22

2. Secondary Outcome: Clinical Status Using CGI-I Score During ON Time
Description: Clinical Global Impression - Global Improvement (CGI-I) is a single-item rating scale used to evaluate a patient's condition relative to baseline on a 7-point scale, regardless of whether the improvement is related to the investigational medicinal product (IMP). The scale ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 16
Population: FAS; last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 151 | 157
units on a scale | 3.56 (0.07) | 3.15 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.61 to -0.22], Standard Error of Mean 0.10

3. Secondary Outcome: Change From Baseline in UPDRS-ADL Score During OFF Time
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worse outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: activities of daily living (ADL) - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
Time Frame: Baseline and Week 16
Population: FAS; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 152 | 158
units on a scale | -1.20 (0.28) | -2.21 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.0075, ANCOVA; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-1.75 to -0.27], Standard Error of Mean 0.37

4. Secondary Outcome: Change From Baseline in UPDRS Motor Score During ON Time
Description: UPDRS is a 42-item rating scale designed to assess Parkinson's Disease-related disability and impairment using a patient interview and a physical examination. It has 4 parts and 4 subsection scores. A higher score indicates a worse outcome. I: mentation, behaviour and mood symptoms - 0 to 16; II: ADL - 0 to 52; III: motor function - 0 to 108; IV: complications of dopaminergic therapy - 0 to 23. Subsection scores for I to III are used to calculate a total score that ranges from 0 (no disability) to 176 (total dependence).
Time Frame: Baseline and Week 16
Population: FAS; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Azilect®
Number analyzed (Participants) | 152 | 158
units on a scale | -1.75 (0.55) | -3.34 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Azilect®; Test type: Superiority or Other; p = 0.0317, ANCOVA; Median Difference (Final Values) = -1.60, 95% CI 2-sided [-3.05 to -0.14], Standard Error of Mean 0.74

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 16-week double-blind treatment period and 4-week safety follow-up period. Other Adverse Events: 16-week double-blind treatment period.
Arm/Group | Placebo | Azilect®
Serious Adverse Events (participants affected / at risk) | 5/158 | 7/163
Other Adverse Events (participants affected / at risk) | 12/158 | 11/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Azilect® (N=163)
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0
Peripheral Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Parkinson's Disease (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Delusional Perception (Psychiatric disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Venous Stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Azilect® (N=163)
Dyskinesia (Nervous system disorders) | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published. Authors of the primary publication based on this study must fulfil the criteria defined by the International Committee of Medical Journal Editors (ICMJE).

The primary publication must be published before any secondary publications are submitted for publication.